CLINICAL TRIAL: NCT01658709
Title: Using Dynamic Postural Control and Functional Testing to Predict Ankle Injury in Adolescent Athletes
Brief Title: Predicting Ankle Injury Through Clinical Functional Measures in Adolescent Athletes
Status: Completed | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Phillip Gribble, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Other Study IDs: UTHSC-15
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Other Instability, Ankle and Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankle Injured: Volunteers with an ankle injury
- Healthy: Healthy Volunteers

SUMMARY:
The objective of this study is to determine if a clinical measure can be used effectively to predict ankle injury in high school and collegiate athletes across a variety of sports.

Hypothesis: For each ankle injury category (lateral ankle sprain, medial ankle sprain, syndesmosis ankle sprain, Achilles rupture, fracture) participants that suffer these injuries will have a significantly lower SEBT normalized composite score and FMS composite score compared to those participants that do not suffer the injury

Hypothesis #1b: Similar to a previous study examining high school basketball players22, using receiver operator characteristic (ROC) curves, we will be able to calculate likelihood ratios, odds ratios, sensitivity and specificity and determine the ideal cut-off point of the SEBT normalized composite score and FMS composite score that will be able to predict the risk of each ankle injury category (lateral ankle sprain, medial ankle sprain, syndesmosis ankle sprain, Achilles rupture, fracture).

Athletes from identified sites will perform measures of the star excursion balance test (SEBT) and the Functional Movement Screen FMS before the first day of practice. During the competition season, the number of practice and competition person exposures, as well as the number of ankle injuries, will be recorded. The rate of ankle injuries/exposure will be calculated and compared with the pre-season SEBT scores to create a simple and a complex prediction model for risk of ankle injury

DETAILED DESCRIPTION:
The objective of this study is to determine if a clinical measure of dynamic postural control, the star excursion balance test (SEBT), and a simple functional testing battery, the Functional Movement Screen (FMS), can be used effectively to predict ankle injury in high school and collegiate athletes across a variety of sports.

Males and females between the ages of 14 and 24 enrolled at one of three designated high schools in Toledo, OH or at the University of Toledo will be recruited for this study. Eligible participants will be signed up and medically cleared to participate in football, basketball, baseball, softball, soccer, volleyball, and/or cross country during the 2012/2013 academic year. Participants will be healthy and must be cleared by a physician for full participation at the time of enrollment in the study. All the enrolled student athletes will be made aware of the study and the requested prior to their pre-season physicals by the coaching staff and ATC prior to the beginning of the first day of practice. Consent and assent will be obtained using appropriate university approved forms. In this prospective study design, pre-season dynamic postural control data and previous injury history will be collected from the high school and collegiate athletes. These athletic facilities are all serviced by certified Athletic Trainers (ATC) and physicians associated with the University of Toledo and the University of Toledo Medical Center. Prior to the beginning of the 2012/2013 competition seasons, athletes from the identified sites will, as part of their pre-season physical exam requirements, perform measures of the SEBT and the FMS before the first day of practice. The performance of the SEBT and the FMS are explained in detail in the attached protocol. During the competition season, the number of practice and competition person exposures, as well as the number of ankle injuries, will be recorded by the ATC at each school. Injury incidence is explained in detail in the attached protocol. At the end of the competition seasons, the rate of ankle injuries/exposure will be calculated and compared with the pre-season SEBT scores to create a simple and a complex prediction model for risk of ankle injury.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Athletes between 14 and 24
* Enrolled in designate area high schools

Exclusion Criteria:

-

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males and female athletes between the ages of 14 and 24 enrolled at one of three designated high schools in Toledo, OH or at the University of Toledo will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gribble, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ankle Injured | Healthy
Started | 59 | 318
Completed | 59 | 318
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle Injured | Healthy | Total
Number analyzed (Participants) | 59 | 318 | 377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 318 | 377
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (2.2) | 15.8 (2.1) | 15.7 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 59 | 318 | 377
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59 | 318 | 377

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Balance: (Star Excursion Balance Test)
Description: The clinical measure of dynamic postural control is represented as a reaching distance normalized to leg length. This is calculated by taking the average liner reaching distance (cm) of the test trials and dividing by the participant's leg length (anterior superior iliac spine to the inferior pole of the medial malleolus of the tibia), also in cm. The resulting ratio is multiplied by 100 and the measure reported as "% of leg length". This value was established in the literature as the standard outcome for reporting Star Excursion Balance Test data.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: % of leg length
Arm/Group | Ankle Injured | Healthy
Number analyzed (Participants) | 59 | 318
% of leg length | 72.3 (8.5) | 78.0 (7.4)

ADVERSE EVENTS:
Arm/Group | Ankle Injured | Healthy
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/318
Other Adverse Events (participants affected / at risk) | 0/59 | 0/318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes